CLINICAL TRIAL: NCT06348771
Title: Postprandial Inflammation and Peanuts in Older Adults
Brief Title: Postprandial Inflammation and Nuts (PIN) in Older Adults
Acronym: PIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Sue A. Shapses, Ph.D., RD, Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Pro2023001579
Record Dates: First submitted 2024-03-22; First posted 2024-04-05 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-01

CONDITIONS: Healthy Aging; Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Fatty Acids, Monounsaturated; Fatty Acids; Meals

STUDY DESIGN:
Intervention Model Description: Higher SFA meal vs higher MUFA (nut) meal in individuals with overweight and obese
Masking Description: No masking but participants are not told which foods in a given meal are higher in one fatty acid or another. 16 will be enrolled as per the sample size calculation for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- saturated fatty acids (SFA) meal (Active Comparator): mixed meal test over 6 hours
  Interventions: Behavioral: monounsaturated fatty acids (MUFA) peanut meal
- monounsaturated fatty acids (MUFA) peanut meal (Experimental): mixed meal test over 6 hours
  Interventions: Behavioral: monounsaturated fatty acids (MUFA) peanut meal

INTERVENTIONS:
Behavioral: monounsaturated fatty acids (MUFA) peanut meal — mixed meal tolerance test and postprandial measurements
  Other Names: Saturated fatty acid (SFA) meal

SUMMARY:
The aging population is rapidly increasing, and it is important to identify dietary factors that can prevent disease and promote health in this group. Legumes, such as peanuts, are a plant-based food high in protein and unsaturated fat making this a healthy choice, but are not consumed frequently enough in older adults. Studies have shown that regular nut consumption is associated with lower adiposity and reduced weight gain and inflammation. Given these findings, this study will examine the postprandial effects of meals with 2 levels of saturated fatty acids (SFA) on metabolic endotoxemia, inflammation and satiety, using a randomized cross-over design. The low SFA meal includes peanuts that are high in monounsaturated fatty acids (MUFA) and this will be compared to a high SFA meal. The results of this study have the potential to provide valuable insights into the role of peanuts in promoting health and preventing disease in at-risk older adults.

DETAILED DESCRIPTION:
The aging population is rapidly increasing, and it is important to identify dietary factors that can prevent disease and promote health in this group. Legumes, such as peanuts, are a plant-based food high in protein and unsaturated fat making this a healthy choice but are not consumed frequently enough in older adults. Studies have shown that regular nut consumption is associated with lower adiposity and reduced weight gain, and several dietary pattern studies indicate that nuts and legumes are associated with better bone health. Given these findings, this study will address the postprandial effects of meals with 2 levels of saturated fatty acids (SFA) on metabolic endotoxemia, inflammation and satiety, using a randomized cross-over design. The low SFA meal includes peanuts that are high in monounsaturated fatty acids (MUFA) and the serum endotoxin (lipopolysaccharide, LPS) postprandial response will be compared to a high SFA meal. Baseline measurements will include body composition and serum lipids and glucose. The objectives of the study are: 1. To determine the endotoxin and inflammatory response to a meal with two levels of saturated fat in older individuals with overweight or obesity using a randomized cross-over design; 2. To evaluate satiety and fullness in response to the two meals. It is hypothesized that postprandial circulating endotoxin and inflammation will be higher, and satiety will be similar after the SFA enriched compared to the lower SFA (peanut based) meal. A sample size analysis indicates that 16 participants are needed (α set at 0.05, and power set at 90%) to detect a significant difference in endotoxin between groups. Assuming a 10% dropout, up to 18 individuals will be enrolled. The results of this study have the potential to provide valuable insights into the role of peanuts in promoting health and preventing disease in at-risk older adults.

ELIGIBILITY:
Inclusion Criteria:

* Older adults across all racial/ethnic groups
* Older men, and postmenopausal women > 2 years since last menses.

Exclusion Criteria:

* Anemia
* Diagnosed with, active, or history of liver cirrhosis, chronic or persisting hepatitis
* Diagnosed with, active, or history of cancer
* History of gastrointestinal disease or surgical procedure for weight loss.
* Diagnosed with immune diseases, type 1 or 2 diabetes, pancreatitis, metabolic bone disease or infectious diseases
* Any surgery in the past 6 months
* Currently using or have used antibiotics continuously > 3 days in the past 3 months
* Regular use of medications for that affect the gastrointestinal tract, cholecystitis, urinary tract infection, significant renal disease, severe organic diseases including coronary heart disease, myocardial infarction, infectious diseases including pulmonary tuberculosis and AIDS
* Known allergy or intolerance to any ingredients in the meal intervention
* Recent colonoscopy (within the previous two months)
* Uncontrolled hypertension or uncontrolled severe hyperlipidemia.
* Participation in another clinical research trial that may interfere with the results of this study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Concentration of Endotoxin | Change over 6 hour MMT
  serum

SECONDARY OUTCOMES:
Concentration of Glucose and Insulin | Change over 6 hour MMT
  serum (mg/dL)
Concentration of Triglyceride | Change over 6 hour MMT
  serum
Appetite | Change over 6 hour MMT
  visual analogue scale from 0 (not at all) to 14 (extremely)
Concentration of Inflammatory markers | Change over 6 hour MMT
  Interleukin-6, tumor necrosis factor-alpha, plasminogen activator inhibitor-1, lipopolysaccharide binding protein, hs-C reactive protein (grams/volume)

OTHER OUTCOMES:
Concentration of zonulin | Baseline only
  serum permeability marker
Lipid Profile | Baseline only
  serum
Characterization of the Microbiome | Baseline only
  alpha and beta diversity of bacteria in feces
Concentration of incretin hormones | Change over 6 hour MMT
  serum GLP-1, gherlin, peptide YY (grams/volume)
Concentration of Bone regulating markers | Fasting and change over 6 hour MMT
  Serum carboxyterminal crosslinking telopeptide of type I collagen (CTX), Procollagen type-I aminoterminal propeptide (PINP), Osteocalcin (grams/volume)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Shapses, PhD, Principal Investigator — Rutgers, the State University of NJ
Locations (2):
- United States (2):
  - Foran Hall, New Brunswick, New Jersey
  - Rutgers University - NJ Inst Food Nutrition & Health, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No
Individual participant data that underlie the results and after deidentification will be shared upon request for researchers who provide a methodologically sound proposal (and IRB approved).

DOCUMENTS (1):
  • Informed Consent Form (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT06348771/ICF_000.pdf